CLINICAL TRIAL: NCT03283969
Title: Probe Study Investigation on the Influence of Freeze Dried Strawberry Consumption on Gut Microbiota, Intestinal Health, Metabolic Phenotype and Cardiovascular Risk in Overweight and Obese Individuals.
Brief Title: Influence of Freeze Dried Strawberry Consumption on Gut Microbiota and Cardiovascular Health.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 956223
Record Dates: First submitted 2017-09-13; First posted 2017-09-15 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2022-06

CONDITIONS: Microbial Colonization; Cardiovascular Diseases; Obesity
MeSH Terms: conditions — Communicable Diseases; Cardiovascular Diseases; Obesity

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, controlled crossover dietary intervention trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: The test powders where pre-packaged by the study sponsor and sent to the investigators coded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Powder (Placebo Comparator): Isocaloric powder
  Interventions: Other: Freeze Dried Strawberry Powder; Other: Isocaloric powder
- Freeze Dried Strawberry Powder (Experimental): Contains freeze dried strawberries
  Interventions: Other: Freeze Dried Strawberry Powder; Other: Isocaloric powder

INTERVENTIONS:
Other: Freeze Dried Strawberry Powder — Study participants will be randomized to receive either the freeze dried strawberry powder or the control powder first. They will be instructed to consume 39g of the powder, mixed in water, every day for 4 weeks.
Other: Isocaloric powder — Isocaloric powder

SUMMARY:
This proposal seeks to build upon studies, including ours, on the favorable effects of California strawberries on vascular health. Freeze dried strawberry powder (FDSP) contains a number of nutrients that may have beneficial effects on plasma lipids and vascular function, as well as on the composition of the gut microbiota; changes in the gut microbiota can in turn have secondary positive effects on the vascular system as well as on other physiological functions that are important determinants of health and disease. The proposed project will seek to determine the influence of short-term FDSP intake on the gut microbiota composition, and select microbial-derived metabolites from stool, serum and urine, and their relationship to microvascular function. Secondary outcomes will include the influence of the FDSP on circulating levels of nitrate and nitrite and trimethylamine oxide (TMAO) as markers of vascular health that are influenced by both dietary intake and the oral and gut microflora, with blood pressure as an additional vascular outcome.

DETAILED DESCRIPTION:
A randomized, double-blind, controlled crossover design will compare the short-term (two and four week) response to FDSP intake compared to an isocaloric control powder in overweight and obese adults. Twenty overweight or obese male or postmenopausal females (40-65 years of age) will be randomized to consume 39 g of FDSP or a control powder for four weeks in a crossover design with a four week washout period. Changes in stool microbial communities and microbial metabolites will be assessed, and examined for their potential influence on microvascular function.

ELIGIBILITY:
Inclusion Criteria:

* Male or postmenopausal female: 40-65 years
* Women: lack of menses for at least two years.
* Subject is willing and able to comply with the study protocols.
* Subject is willing to participate in all study procedures
* BMI 25.0 - 35 kg/m2

Exclusion Criteria:

* BMI ≥ 35 kg/m2
* Dislike or allergy for strawberries or strawberry products
* Self-reported use of daily anticoagulation agents including aspirin, NSAIDs
* Vegan, Vegetarians, food faddists or those consuming a non-traditional diet
* Fruit consumption ≥ 2 cups/day
* Regular consumption of strawberries (2-3 cups/week)
* Vegetable consumption ≥ 3 cups/day for females
* Fatty Fish ≥ 3 times/week
* Coffee/tea ≥ 3 cups/day
* Dark chocolate ≥ 3 oz/day
* Self-reported restriction of physical activity due to a chronic health condition
* Self-reported chronic/routine high intensity exercise
* Self-reported diabetes
* Blood pressure ≥ 140/90 mm Hg
* Self-reported renal or liver disease
* Self-reported heart disease, which includes cardiovascular events and stroke
* Inability to properly place or wear the PAT probes or abnormal measurements on pre- screening PAT
* Abnormal Metabolic or CBC panels (laboratory values outside the reference range) if determined to be clinically significant by the study physician.
* Self-reported cancer within past 5 years
* Self-reported malabsorption
* Currently taking prescription drugs or supplements.
* Use of multi-vitamin and mineral other than a general formula of vitamins and minerals that meet the RDA
* Not willing to stop any supplement use, including herbal, plant or botanical, fish oil, oil supplements a month prior to study enrollment.
* Indications of substance or alcohol abuse within the last 3 years
* Screening LDL ≥ 190 mg/dl for those who have 0-1 major risk factors apart from LDL cholesterol (i.e. family history of premature coronary artery disease (male first degree relative < 55 years; CHD in female first degree relative < 65 years), cigarette smoker, HDL-C ≤ 40 mg/dL].
* Screening LDL ≥ 160 mg/dl for those who have 2 major risk factors apart from LDL cholesterol [i.e. family history of premature coronary artery disease (male first degree relative < 55 years; CHD in female first degree relative < 65 years), cigarette smoker, HDL-C ≤ 40 mg/dL]. (using NCEP calculator http://cvdrisk.nhlbi.nih.gov/calculator.asp);
* Screening LDL ≥ 130 mg/dl for those who have 2 major risk factors apart from LDL cholesterol [i.e. family history of premature coronary artery disease (male first degree relative < 55 years; CHD in female first degree relative < 65 years), cigarette smoker, HDL-C ≤ 40 mg/dL], and a Framingham 10-year Risk Score 10-20% (using NCEP calculator http://cvdrisk.nhlbi.nih.gov/calculator.asp).
* Current enrollee in a clinical research study.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Peripheral Arterial Tonometry (PAT) | 10 weeks
  microvascular function testing

SECONDARY OUTCOMES:
Gut Microbiome | 10 weeks
  assessment of gut microbial populations
Untargeted Metabolomics | 10 weeks
  assessment of primary metabolites
Plasma Cholesterol | 10 weeks
  plasma cholesterol
Plasma LDL | 10 weeks
  LDL
Plasma HDL | 10 weeks
  HDL
Nitrate | 10 weeks
  Circulating levels of Nitrate
Nitrite | 10 weeks
  Circulating levels of Nitrite

CONTACTS AND LOCATIONS:
Overall Officials: Carl L Keen, PhD, Principal Investigator — University of California, Davis
Locations (1):
- University of California, Davis; Department of Nutrition, Davis, California, United States

IPD SHARING:
Plan to Share IPD: No